CLINICAL TRIAL: NCT06652113
Title: The Efficacy of Hydroxychloroquine Combined With Levothyroxine in Euthyroid Women With Thyroid Antibody Positive and Unexplained Recurrent Pregnancy Loss：A Multicenter, Randomized Controlled Study
Brief Title: Effect of HCQ Combined With LT4 on LBR in Euthyroid Women With URPL and TPO-Ab
Acronym: QT-LIFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-342-01
Record Dates: First submitted 2024-06-25; First posted 2024-10-22 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Pregnancy Loss; Euthyroid With Thyroid Antibodies
Keywords: live birth; euthyroid; thyroid peroxidase antibody; recurrent pregnancy loss
MeSH Terms: interventions — Hydroxychloroquine; Thyroxine

STUDY DESIGN:
Intervention Model Description: open-labeled multicenter randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hydroxychloroquine and levothyroxine group (Experimental): Corresponding oral treatment will be initiated after randomization and preconceptually, and continue to the end of pregnancy or until 60 weeks post-randomisation if pregnancy does not occur. Patients in the experimental group will be given a combined oral treatment of hydroxychloroquine (HCQ) and levothyroxine. Hydroxychloroquine sulfate tablets (Fenle, 0.1g) will be given at a total daily dose of 0.2g to 0.4g based on individual weight: patients weighing ≤46kg take HCQ tablets 0.2g/d, patients weighing >46kg and <62kg take HCQ tablets 0.3g/d, patients weighing ≥62kg take HCQ tablets 0.4g/d. Levothyroxine sodium tablets (Euthyrox, 50 μg) will be given 12.5μg ~50 μg daily based on patients' TSH levels and weights: TSH ≥ 2.5 mIU/L, the dosage is 50 μg/d; TSH < 2.5 mIU/L, the dosage is 25 μg/d; when the patient's weight is less than 50kg, the dosage is reduced by 50%.
  Interventions: Drug: hydroxychloroquine and levothyroxine
- levothyroxine group (Other): Corresponding oral treatment will be initiated after randomization and preconceptually, and continued to the end of any pregnancy or until 60 weeks post-randomisation if pregnancy does not occur. Patients assigned in the control group will be given levothyroxine daily. Levothyroxine sodium tablets (Euthyrox, 50 μg) will be given 12.5μg ~50 μg daily based on patients' TSH levels and weights: TSH ≥ 2.5 mIU/L, the dosage is 50 μg/d; TSH < 2.5 mIU/L, the dosage is 25 μg/d; when the patient's weight is less than 50kg, the dosage is reduced by 50%.
  Interventions: Drug: Levothyroxine

INTERVENTIONS:
Drug: hydroxychloroquine and levothyroxine — Hydroxychloroquine sulfate tablets (Fenle, 0.1g) will be given at a total daily dose of 0.2g to 0.4g based on individual weight as described above. During the study, if TSH is higher than 4.0 mIU/L or exceeds the lower limit of the reference range of the center in the first trimester, or TSH level exceeds the normal range of the center during the second or the third trimester, subjects will be instructed to suspend the medication and visit the Department of Endocrinology.
  Arms: hydroxychloroquine and levothyroxine group
Drug: Levothyroxine — Levothyroxine sodium tablets (Euthyrox, 50 μg) will be given 12.5μg ~50 μg daily based on patients' TSH levels and weights as described above. During the study, if TSH is higher than 4.0 mIU/L or exceeds the lower limit of the reference range of the center in the first trimester, or TSH level exceeds the normal range of the center during the second or the third trimester, subjects will be instructed to suspend the medication and visit the Department of Endocrinology.
  Arms: levothyroxine group

SUMMARY:
The goal of this clinical trial is to learn if combined treatment of levothyroxine and hydroxychloroquine would improve the live birth of euthyroid women with thyroid peroxidase antibodies and unexplained recurrent pregnancy loss.

Researchers will compare combined treatment of levothyroxine and hydroxychloroquine to a treatment of levothyroxine alone to see if combined treatment works to improve live birth of euthyroid participants with thyroid peroxidase antibodies and unexplained recurrent pregnancy loss.

Participants will:

* Receive combined treatment of levothyroxine and hydroxychloroquine or treatment of levothyroxine alone every day at least 8 weeks before pregnancy, and continue their treatment till the end of pregnancy.
* Visit the clinic 4 weeks and 8 weeks after their treatments, and every 12 weeks before they get pregnant for checkups and tests. During their pregnancy, they will visit the clinic before gestation of 12 weeks, and will be followed up with phone call in the second trimester and after parturition.

DETAILED DESCRIPTION:
Thyroid peroxidase antibodies (TPO-Ab) in euthyroid women are associated with recurrent pregnancy loss. According to 2017 Guidelines of the American Thyroid Association, administration of levothyroxine (LT4) to TPO-Ab-positive euthyroid pregnant women with a prior history of loss may be considered given its potential benefits in comparison with its minimal risk. However, it is a weak recommendation with low-quality evidence. Recently published randomised clinical trials showed that administration of LT4 does not improve pregnancy outcomes of euthyroid thyroid peroxidase antibody positive women with recurrent pregnancy loss. Published data showed TPO-Ab is related to immune imbalance. Hydroxychloroquine is a widely used immune modulator even in fields of autoimmune disorders during pregnancy and lactation. Nevertheless, the effect of hydroxychloroquine combined with LT4 on live birth rate of euthyroid women with TPO-Ab and unexplained recurrent pregnancy loss is unclear. Therefore, we designed a multicenter RCT to verify the study hypothesis that combined treatment of levothyroxine and hydroxychloroquine would improve the live birth rate of euthyroid women with thyroid peroxidase antibodies and unexplained recurrent pregnancy loss.

ELIGIBILITY:
Inclusion criteria:

1. Women with history of two or more pregnancy loss with the same male partner (including biochemical pregnancies).
2. Karyotype analyses show no pathological abnormalities in each individual of the recruited couple.
3. Women aged between 20 and 40 years old (including 20 and 40).
4. Lupus anticoagulant (LA), anticardiolipin antibody (ACA), and anti-beta2-glycoprotein I antibodies (anti-β2-GP1 Ab) tests are all negative.
5. It is confirmed by ultrasound or hysteroscopy that there are no pathological lesions that affect the morphology of the uterine cavity (such as submucosal uterine fibroids, uterine malformations).
6. TPO-Ab positive (TPO-Ab > 60 IU/mL using the Siemens kit of electrochemiluminescence method, or TPO-Ab > 34 IU/mL using the Roche kit of chemiluminescence method).
7. Biochemically euthyroid. TSH, free triiodothyronine (FT3), and free thyroxine (T4) are all within the reference range of corresponding laboratory testing in each research center.

Exclusion criteria:

1. Rheumatic diseases, such as systemic lupus erythematosus, undifferentiated connective tissue disease, etc.
2. Metabolic or endocrine diseases, such as diabetes.
3. Abnormal renal function: plasma creatinine level ≥130 μmol/L or abnormal liver function: alanine aminotransferase ≥80U/L or aspartate aminotransferase ≥80U/L.
4. Hypertension and malignant tumors.
5. Under treatment with glucocorticoids or immunosuppressor, including cyclosporine, azathioprine, prednisone, and methylprednisolone.
6. Body Mass Index (BMI) >28kg/m2.
7. Past history of hyperthyroidism, hypothyroidism, and thyroid malignant tumors;
8. Allergy to 4-aminoquinoline compound, or those with retinal or visual field lesions caused by 4-aminoquinoline compound.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 796 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2035-03 (Estimated); Study Completion 2037-03 (Estimated)

PRIMARY OUTCOMES:
Birth of a living child beyond 28 weeks | After birth, within 24 months after randomization
  The primary outcome is the proportion of women with a live birth at or beyond 28 completed weeks. This proportion will be calculated with the denominator totalling all women randomised, and the numerator (i.e., treatment successes) totalling women who conceive within 60 weeks of randomisation and go on to give live birth at or beyond 28 weeks gestation.

SECONDARY OUTCOMES:
Clinical pregnancy at 5 to 8 weeks | At 5-8 weeks of pregnancy
  It is the proportion of women with a cardiac activity confirmed by ultrasound during 5 to 8 weeks of gestation. This proportion will be calculated with the denominator totalling all women randomised, and the numerator totalling women who have clinical pregnancy within 60 weeks of randomisation.
Miscarriage <28 weeks | At 28 weeks of pregnancy
  Miscarriage that occurs less than 28 weeks of gestation
Gestation at miscarriage, weeks | After the time of miscarriage, within 24 months after eligibility
  Gestation at miscarriage, weeks
On-going pregnancy at 12 weeks | At 12 weeks of pregnancy
  On-going pregnancy at 12 weeks
Gestation at delivery >34 weeks/>37 weeks | After birth, within 24 months after eligibility
  Number of women who have a delivery at least 34 weeks of gestation. Number of women who have a delivery at least 37 weeks of gestation.
Gestation at delivery, weeks | After birth, within 24 months after eligibility
  Gestation at delivery, weeks
Birth weight, grams | At birth, within 24 months after eligibility
  Birth weight, grams
APGAR score at 1 minute/5 minutes | After birth, within 24 months after eligibility
  APGAR score at 1 minute/5 minutes of the neonates.
birth defects | At or short after birth, within 24 months after eligibility
  Birth defects of the neonates.
Maternal antenatal complications,intrapartum complications,maternal postnatal complications | up to birth/immediately after delivery
  Hypertensive disorders of pregnancy, gestational diabetes, placenta previa, placental abruption, polyhydramnios, oligohydramnios, fetal growth restriction, postpartum hemorrhage and so on.
Time to pregnancy. | At 5-8 weeks of pregnancy
  It refers to the time interval from patients trying to prepare for pregnancy (after 8 weeks of medication) to successful pregnancy (intrauterine pregnancy confirmed by ultrasound).
live birth rate after at least 28 weeks of gestation among pregnant patients | After birth, within 24 months after randomization
  It is the proportion of women with a live birth at or beyond 28 of completed weeks. This proportion will be calculated with the denominator totalling all women who have clinical pregnancy within 60 weeks of randomisation, and the numerator totalling women who have a live birth at or beyond 28 of completed weeks.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong